CLINICAL TRIAL: NCT06395623
Title: Study of Acupoints in Diminished Ovarian Reserve Based on Biological Characteristics：A Case-control Study
Brief Title: Study of Acupoints in Diminished Ovarian Reserve Based on Biological Characteristics
Status: Recruiting | Type: Observational
Sponsor: Xiaomei Shao (Other)
Collaborators: Hangzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 2022YFC3500401
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Diminished Ovarian Reserve
Keywords: Biological Characteristics; Acupoint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with DOR: 50 patients diagnosed with DOR will be recruited in this group to get detectionsof pain threshold, infrared thermal image, resistance, micro-circulation, and biological ultra-weak luminescence at the relevant body surface areas and meridian acupoints and the blood test of serum FSH(follicle-stimulating hormone) and AMH(Anti-Müllerian Hormone).
- Healthy participants: 50 healthy participants in this group will achieve the same detections of biological characteristics and blood test as well.

SUMMARY:
Diminished Ovarian Reserve (DOR) is characterized by decreased female fertility, menstrual disorders and perimenopausal symptoms due to sex hormone deficiency or fluctuations. For now, there are no uniform diagnostic criteria or an ideal single detection index for DOR because of its insidious etiology and pathogenesis,theories suggest that there are specific changes in the body surface or acupuncture points in a pathological state. By detecting the biological characteristics of relevant meridian points and exploring the specificity and regularity of it.

DETAILED DESCRIPTION:
There will be a multi-center, case-control, observational experiment. 50 patients with DOR and 50 healthy participants will be involved from Third Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou TCM Hospital Affiliated to Zhejiang Chinese Medicine University and social recruitment. Modern instruments are used to regularly test the pain threshold, infrared thermal image, resistance, micro-circulation, and biological ultra-weak luminescence. There will be no randomized methods and blindness for subjects, while assessors and statisticians are masked from patients or healthy people. The study is aim to explore the the relevance between meridian acupoints and DOR.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patient with DOR:

* 18 years old ≤ age < 40 years old, female;
* Clinical diagnosis of Diminished Ovarian Reserve: meet both items in twice tests with an interval of at least 4 weeks(tested between 2rd to 4th day of menstrual cycle):

  1. 10 IU/L < FSH < 20 IU/L,
  2. Anti-Müllerian hormone(AMH) < 1.1ng/mL.
* without any mind disease, willing to participate in the study and sign the informed consent.
* without any other treatment.

Inclusion criteria for healthy participants:

* healthy participants who can provide medical examination reports within the past 1 year and have routine physical examination conducted by researchers to confirm that there are no serious underlying diseases of the reproductive system, urinary system, blood, endocrine, nervous system, etc.;
* without symptoms of oligomenorrhea or amenorrhea at present;
* between the ages of 18 to 40, female;
* without any mind disease, volunteering to participate in the study and sign the informed consent.

Exclusion Criteria:

Exclusion Criteria for patient with DOR

* Low or no response to exogenous gonadotropins, or with congenital anomalies in the development of the reproductive tract;
* Pregnant or breastfeeding;
* Abnormal body temperatures at the moment;
* Psychopath, alcoholic, Patient with severe depression, history of substance abuse and severe primary diseases of cardiovascular, liver, kidney and hematopoietic system;
* Currently enrolled in other clinical trials or refuse to cooperate with the study protocol.

Exclusion Criteria for healthy participants

* Patient with mental illness, severe depression, alcohol dependence or a history of drug abuse;
* In pregnant or breastfeeding;
* abnormal body temperature at present;
* Participants who are currently participating in other clinical trials or who do not cooperate with the study protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study targets at patients with DOR and healthy participants. The diagnostic criteria of DOR were based on<Consensus on Cinical Diagnosis and Management of Diminished Ovarian Reserve(2022)> and <Obstetrics and Gynecology(9th edition)>
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Temperature of acupoint by infrared thermal image | baseline
  Infrared thermography (The NEC R550 infrared thermal imager and the InfRec Analyzer NS9500 computer software) will be used to measured the temperature of the meridian acupoints. The measurements are taken at participants' follicular phase.
Pain threshold | baseline
  Pain threshold of related acupoints will be tested by pressure pain threshold gauge (PTG). Assessors will put continuous pressure on the surface of acupoints vertically until participants feel pain to measure the threshold.

SECONDARY OUTCOMES:
Serum follicle-stimulating hormone (FSH) | baseline
  The increasing of FSH is widely clinical accepted for measuring ovarian function, which is one of the main symptoms of Diminished Ovarian Reserve. Participants in this study will be asked to take the serum FSH text between day2 to day4 of menstrual period in whole observation.
Serum Anti-Müllerian Hormone (AMH) | baseline
  AMH is another recommend index to measure ovarian function. Compared to FSH, Anti-Müllerian Hormone has less fluctuation and more accuracy. The normal value of serum AMH is 2-6.8ng/ml in follicular phase, and lower the value, the worse condition. The serum AMH will be measured on day 2-4 of the menstrual cycle at the basement and the end of the treatment.
The modified Kupperman Index(KI) | baseline
  The modified Kupperman Index (KI) is widely used for female self-evaluation of the severity of menopausal symptoms in clinical practice. It values 13 items of menopausal symptoms on a scale of 0 to 3. The final score of KI is the sum of each score multiplied with the base score respectively, ranging from 0-63. The final KI score is less than 6 means normal, between 6 to 15 are classified as mild, 16 to 30 as moderate, and greater than 30 as severe.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China